CLINICAL TRIAL: NCT00333593
Title: Randomized, Cross Over Study Comparing Standard Hemodialysis to Hemodialysis With a Novel Polyamide Membrane (P2SH) in Patients With Sepsis and Acute Renal Failure
Brief Title: Super High-Flux - High Volume Dialysis in Sepsis-Induced Acute Renal Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H2003/01440
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Sepsis; Acute Renal Failure
Keywords: Dialysis; Large pore dialyser; Cytokines; Noradrenaline
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

INTERVENTIONS:
Device: Large pore dialyser
Device: Standard dialyser

SUMMARY:
Patients within the intensive care unit who have severe infections causing shock and kidney failure have almost a 60% risk of dying despite antibiotic therapy, surgical drainage of the site of infection and intensive care support with fluids, nutrition, mechanical ventilation and continuous artificial kidney support. This persistently high death rate continues to stimulate the development of new approaches to the treatment of septic shock.

Much clinical and molecular biology research suggests that these patients die because of an uncontrolled immune system's response to infection. This response involves the production of several substances (so called "humoral mediators"), which enter the blood stream and affect the patient's organs ability to function and the patient's ability to kill germs. These substances may potentially be removed by new artificial filters similar to those currently used during continuous hemofiltration (the type of artificial kidney support used in intensive care).

Recent investigations by ourselves and others, however, have made the following findings:

1. Standard filters currently used in intensive care are ineffective in removing large amounts of these "humoral mediators" because the holes in the filter are too small to allow all of them to pass through
2. The standard filters currently used in intensive care are also ineffective in removing large amounts of these "humoral mediators" because the standard filtration flow through the membrane is less than 100 ml/min
3. When the filtration flow through the membrane is increased to above 100ml/min, patients require a lesser dose of drugs to support their blood pressure which is an indirect sign that the filters are clearing some of the "humoral mediators"
4. Even when the blood flow through standard filters is increased to above 100ml/min, there is still not optimal clearing of "humoral mediators" It is possible, however, that, using a different filter membrane with bigger holes in it, would make it easier to clear the blood of these "humoral mediators". It is thought that this would be noticeable clinically in the amount of drugs required to support blood pressure.

A filter that has these bigger holes is now available. It is made of the same material as the standard filters that are currently used in the intensive care unit, only the holes have been made bigger to allow these "humoral mediators" to be removed from the blood. This polyamide filter is made of synthetic semipermeable material. This material is highly compatible with human blood. This modified polyamide filter is made of exactly the same compatible material but the holes in the material are slightly larger through a minor modification of the manufacturing process.

This larger hole filter has now been used in preliminary studies in humans and has been found to reduce the blood levels of some "humoral mediators". Laboratory studies conducted by ourselves showed that this new filter can achieve the highest reported clearance of some of the "humoral mediators" with minimal effect on useful proteins in blood such as albumin during hemodialysis. This loss is very small and unlikely to contribute to any detectable clinical changes.

We, therefore, now propose to study the effect of using new large hole filters with hemodialysis in patients with severe infections and acute kidney failure.

We wish to compare the effect of this new therapy to that of standard filters. The new therapy will be considered to be effective if it lowers the amount of drugs used to support blood pressure and if it lowers the blood levels of some "humoral mediators" more than standard therapy. We will also monitor blood levels of important components of blood such as albumin and electrolytes in each group.

This is a pilot study involving only 10 patients who will each receive 4 hours of the standard therapy and 4 hours of the new therapy. Which treatment the patient receives first will be random (like the tossing of a coin). Blood samples will be taken at the start and after 4 hours of each treatment. The waste product of dialysis called spent dialysate will also be collected for the measurement of humoral mediators at the start and after 4 hours of each treatment. The changes in blood pressure and drugs used to support it will be recorded hourly. As patients involved in the study would normally receive hemofiltration because of their kidney failure, all the risks and benefits associated with the procedure would be unchanged. The only risk to patients would come from exposure to a modified membrane and from having two additional spoonfuls of blood taken.

If this new membrane were found to have a major effect on the blood level of "humoral mediators" and on the patients' blood pressure, further studies would then be justified to assess its clinical effects (time in ICU, time in hospital, time on ventilator, duration of organ failure, etc).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The combination of acute renal failure (ARF) and sepsis is associated with a very high morbidity and mortality (1). Accordingly, there have many attempts to develop better treatments for this condition.

Much clinical and molecular biology research suggests that septic shock occurs because of the uncontrolled immune system's response to infection (2-13). This response involves the production of several substances (so called "humoral mediators"), which enter the blood stream and, at different times in the course of the patients' illness, cause either severe inflammation or profound depression of the immune system's ability to kill microbes.

The vast majority of these substances (cytokines, complement anaphylatoxins, platelet activating factor, leukotrienes, chemokines), which are responsible for this state of "blood poisoning" are water soluble and of small to middle molecular weight (up to 40 kilodaltons). These properties make them potentially removal by artificial membranes similar to those used during continuous hemofiltration (the type of artificial kidney support used in intensive care).

It is possible that using a different and more porous membrane, the removal of such cytokines would be much more efficient and the clinical benefits of blood purification would, therefore, be greater.

A membrane of this kind is now available. It is a modification (moderate increase in pore size) of standard material called polyamide, which has already been used in millions of people for dialysis and hemofiltration.

This larger pore polyamide membrane has now been used in preliminary studies in humans (14) and has been found to be capable of lowering the blood levels of a marker cytokine (interleukin-6, molecular weight: 26.2 kD).

In laboratory studies conducted by ourselves, this new polyamide membrane achieves the highest reported cytokine and beta2-Microglobulin - as another marker of removal of middle molecules - clearances in the literature and is associated with a negligible loss of albumin (15).

Recent investigations by ourselves and others, however, have made the following findings:

1. Standard membranes are of only limited effectiveness in filtering these "humoral mediators" (16)
2. Unless high volume plasma-water exchange is applied (100 ml/min), the effect of blood purification on the blood levels of these mediators are minimal (17-20)
3. High volume hemofiltration with standard membranes, results in an improvement in the state of the circulation such that the infusion of drugs used to support blood pressure (noradrenaline) can be decreased (20).
4. Even with high volume hemofiltration the removal of "humoral mediators" such as cytokines is still of limited efficiency (20)

It is possible that using a different and more porous membrane, the removal of such cytokines would be much more efficient and the clinical benefits of blood purification would, therefore, be greater.

A membrane of this kind is now available. It is a modification (moderate increase in pore size) of standard material called polyamide, which has already been used in millions of people for dialysis and hemofiltration.

We, therefore, propose to study the effect of combining hemodialysis and this new polyamide membrane with larger pores in the treatment of patients with sepsis and acute kidney failure. We wish to compare the effect of this new therapy to that of hemodialysis with a standard membrane.

The terms of comparison (outcome measures) will be:

A). The effect of each therapy on the blood concentration of several cytokines (TNF-alpha, IL-1 beta, Il-6, IL-8, and IL-10).

B). The effect of each therapy on the blood concentration of beta2-Microglobulin as another marker of removal of middle molecules.

C). The effect of each therapy on blood pressure and the need for noradrenaline infusion

and, for safety assessment

D). The effect of each therapy on the blood concentration of albumin and electrolytes

If this new membrane were found to have a major effect on the blood concentration of cytokines and on the patients' blood pressure, further studies would then be justified to assess its clinical effects (time in ICU, time in hospital, time on ventilator, duration of organ failure, etc) in further trial.

STUDY OBJECTIVE

The aim of the study is to compare the effect of hemodialysis combined with a larger pore membrane to that of hemodialysis with a standard membrane on

1. the serum concentration of several cytokines (efficacy assessment)
2. the serum concentration and clearance rates of beta2- Microglobulin (efficacy assessment)
3. blood pressure and noradrenaline requirements (efficacy assessment)
4. the serum concentration of albumin and electrolytes (safety assessment)

   NULL HYPOTHESIS

   The use of hemodialysis combined with a larger pore membrane has no effect on serum cytokine or beta2-Microglobulin levels, blood pressure and noradrenaline requirements when compared to hemodialysis with a standard membrane.

   STUDY DESIGN

   This study is a phase I/II equivalent investigation. It is a pilot, randomised, crossover, controlled study. Eligible patients will receive both treatments. However, the order of treatment (first treatment A and then B or vice versa) will be allocated in a random fashion (computer generated random numbers).

   After completing the first treatment, patients will then be crossed over to the alternative treatment.

   Treatments will consist of either:

   A) hemodialysis with a new polyamide (P2SH) membrane for 4 hours or B) hemodialysis with a standard polyamide membrane

   Blood will be sampled (serum cytokine and beta2-Microglobulin measurement) at the start of each treatment and after 4 hours of each treatment. Dialysate will also be collected for the measurement of cytokines and beta2-Microglobulin in order to calculate cytokine and beta2-Microglobulin clearance.

   The changes in blood pressure and noradrenaline dose will be recorded hourly as is routine in Intensive Care. Patient treatment will otherwise continue according to clinical needs and to standard ICU care.

   It is important to note that patients involved in the study would normally receive standard hemofiltration anyway because of their kidney failure, with all the risks and benefits associated with the procedure (insertion of double lumen catheter, extracorporeal circulation, anticoagulation).

   As part of the study, however, they will also receive increased intensity of treatment, 4 hours of exposure to a modified membrane and some additional blood sampling (one spoonful).

   It is possible that the effect of the first therapy would cross over to the second. To control for this crossover effect, statistical comparison will be undertaken according to order of treatment as well as type of treatment, as recently published. (23)

   STUDY POPULATION

   All patients who fulfil the consensus criteria for sepsis (21) and recently proposed criteria for severe ARF (1) are eligible for the study.

   SPECIFIC EXCLUSIONS
   * Patients under 18 years of age.
   * Patients who are pregnant or breastfeeding
   * Patients with a known allergy to polyamide
   * Patients expected to die within 24 hours
   * Patients in whom there are limitations on the intensity of therapy

   ENROLMENT

   Once patient eligibility is established informed consent will be sought from the next of kin. If informed consent is obtained, the patient will be enrolled in the study. The ICU research nurse will be responsible for enrolment and subsequent data collection.

   STUDY PROTOCOL

   Following enrolment and randomisation, the patient will be allocated to either treatment A or B.

   An extracorporeal circuit will be set up for dialysis with the Fresenius 2008 machine.

   The only difference will be that, one filter which is being applied, will be a larger pore polyamide filter. The other filter whic is being applied, will be a standard polyamide filter.

   Each treatment will be applied for 4 hours. After each treatment, the extracorporeal circuit will be flushed with Hartmann's solution and the membrane changed to the alternative material (cross over).

   For each treatment, the following technical settings will apply:
   1. Blood flow at 200 ml/min
   2. Dialysate flow at 300 ml/min
   3. Anticoagulation of filter with prefilter heparin, if necessary (e.g. 1,000 IU/hr)
   4. Bicarbonate-buffered dialysate

   After the completion of the 2 periods of 4 hours of hemodialysis, patients will revert to standard therapy (hemofiltration with AN 69 membrane at 2 L/hr of plasma water exchange) and continue their normal treatment.

   Randomisation and Concealment

   The randomisation will be based on random numbers generated by computer. The allocation to either treatment A or B as the first treatment will be placed in an opaque envelope by an independent person.

   Once consent is obtained, the envelope will be opened and treatment initiated. Filters will be blinded and both will have identical appearance, outlining only "Filter A" or "Filter B", respectively, on a label sticking to each filter.

   For reasons of patient safety, filter monitoring for membrane clotting requires that the filter be visualized at all times.

   EXPECTED SIZE OF TREATMENT DIFFERENCE

   This study is designed to detect a 30% decrease in IL-6 levels. From a previous very similar investigation (19), we also assume a standard deviation equal in size to the effect being tested for. Using non-parametric paired comparison statistics (Wilcoxon ranked sign test), a sample of 10 patients would offer a > 80% power of detecting a 30% difference at an alpha of 0.05 (22).

   CLINICAL OUTCOMES AND DATA ANALYSIS

   Primary analysis will be performed on the basis of intention to treat. Secondary analysis will be performed on per protocol analysis. The primary outcome measure for this study is the clearance and the change in IL-6 levels The secondary outcome is the the clearance and change in the levels of other cytokines and beta2-Microglobulin.

   The other secondary outcome is the change in noradrenaline dose required to maintain baseline mean blood pressure (typically 70 mmHg)

   Treatment groups will be analysed for differences in IL-6 levels after 4 hours of treatment.

   It is expected from clinical observation that the criteria for normal distribution will be violated. Therefore comparison will be performed using a non-parametric test (Wilcoxon ranked sign test). Statistical significance will be set at p<0.05.

   The groups will also be tested for differences in secondary outcome variables. Such secondary outcome variables are:
   1. Absolute change in all serum cytokine levels for each cytokine and for beta2-Microglobulin
   2. Percentage change in noradrenaline dose
   3. Change in blood pressure from pre-treatment value to value after 4 hours of treatment
   4. Percentage change in serum cytokine levels for each cytokine

   Using the primary outcome variable, this study has an 80% power of detecting a 30% difference at an alpha of <0.05.

   It is expected from clinical observation that recruitment of 10 patients will take 3 months.

   Data Collection

   Data collection will be by the Intensive Care Dept. research nurse and research fellows.

   The following variables will be obtained:

   Name, gender, age and medical record number

   Date of admission to ICU

   Admission diagnosis

   SAPS II illness severity score on admission

   Time of onset of septic shock

   Time of onset of ARF

   Time of onset of hemofiltration

   Hemodynamic indices, temperature and biochemical indices at baseline and after 4 hours

   Use of inotropic drugs and dose

   Use of vasopressor drugs and dose

   Hourly urine output (if present)

   Time of onset of mechanical ventilation

   Fluid balance during each 4 hours of treatment

   Albumin and electrolytes at baseline and after 4 hours

   CONCOMITANT MEDICATIONS

   Concomitant medications will be administered according to standard intensive care

   ADVERSE EVENTS

   If any adverse events occur which may be related to the trial device, treatment will be stopped. The event will be immediately reported to the Ethics Committee according to institutional protocol.

   PROTOCOL VIOLATIONS

   All protocol violations will be recorded. It will then be decided whether the nature of such violations has been such that the patient should be excluded from primary data analysis.

   WITHDRAWAL

   The treating clinician will have the right to withdraw the patient from the study if he or she believes that continued participation is jeopardizing the patient's well being.

   Patients who require take back to theatre during the study period for a surgical emergency will be withdrawn from the trial.

   CONSENT TO TRIAL ENROLMENT

   In all patients it may be necessary to ask for consent from the next of kin. All of these patients are mechanically ventilated and too ill to give informed consent

   ETHICAL ISSUES

   The polyamide material used for the study membrane is very safe and has been used in millions of patients. Its modification is exclusively to the pore size, not to its composition. The effect of pore size on protein losses appears minimal for proteins > 60 kD in molecular weight such as albumin. Accurate in vitro testing confirms this.

   Preliminary phase I data also confirms such safety. We consider the potential benefit of this intervention theoretically significant.

   Given the balance of benefits and risks, we consider it ethical to proceed and seek informed consent.

   References
   1. Bellomo R, Ronco C, Kellum JA. Acute renal failure: time for consensus. Intensive Care Med 2001; 27: 1685-1688
   2. Bellomo R, Baldwin I, Ronco C. Rationale for extracorporeal blood purification therapies in sepsis Current Opinion in Critical Care 2000; 6:446-450
   3. Camussi G, Montrucchio G, Diminioni L, Dionigi R. Septic shock: the unravelling of molecular mechanism. Nephrol Dial Transplant 1995; 10:1808-13.
   4. Glauser MP, Zanetti G, Baumgartner JD, Cohen J. Septic shock: pathogenesis. Lancet 1991; 338: 732-736.
   5. Munoz C, Carlet J, Fitting C, Misset B, Bleriot JP, Cavaillon JM. Dysregulation of in vitro cytokine production by monocytes during sepsis. J Clin Invest 1991; 88: 1747-1754.
   6. Randow F, Syrbe V, Meisel C, Krausch D, Zuckerman H, Platzer C, Volk HD. Mechanism of endotoxin desensitization: involvement of interleukin-10 and transforming growth factor. J Exp Med 1995; 181: 1887-1892.
   7. Brandtzaeg P, Osnes L, Ovstebo R, Joo GB, Westvik AB, Kierulf P. Net inflammatory capacity of human septic shock plasma evaluated by a monocyte-based target cell assay: identification of interleukin-10 as a major functional deactivator of human monocytes. J Exp Med 1996 Jul 1;184(1):51-60.
   8. Wolk K, Doecke W, von Baehr V, Volk H, Savat R. Comparison of monocyte functions after LPS- or IL-10- induced re-orientation: importance in clinical immunoparalysis. Pathobiology 1999; 67(5-6): 253-6.
   9. Bone RC, Grodzin CJ, Balk RA. Sepsis: a new hypothesis for pathogenesis of the disease process. Chest 1997;112: 235-43.
   10. Manjuck J, Saha DC, Astiz M, Eales LJ, Rackow EC. Decreased response to recall antigens is associated with deprived co-stimulatory receptor expression in septic critically ill patients. J Lab Clin Med 2000; 135(2): 153-60.
   11. Weighardt H, Heidecke CD, Emmanuilidis K, Maier S, Bartels H, Siewert JR, Holzmann B. Sepsis after major visceral surgery is associated with sustained and interferon-gamma-resistant defects of monocyte cytokine production. Surgery 2000; 127(3): 309-315.
   12. Nerad J, Griffiths JK, Van der Meer JWM, Endres S, Poutsiaka, DD, Keusch GT, Bennish M, Salam, MA, Dinarello CA, Cannon JG. Interleukin-1 (IL-1), IL-1 receptor antagonist, and TNF production in whole blood. J Leuk Biol 1992.;52: 687-92.
   13. Haupt W, Zirngibl H, Stehr A, Riese J, Holzheimer RG, Hohenberger W. Tumor necrosis factor and interleukin-10 production in septic patients and the regulatory effect of plasma. Eur J Surgery 1999; 165(2): 95-10
   14. Morgera s, Buder W, Lehman C, et al. High cut off membrane hemofiltration in septic patients with multiorgan failure. A preliminary report. Blood Purif 2000; 18: 73 (abstract)
   15. Uchino S, Bellomo R, Goldsmith D, Davenport P,Cole L, Baldwin I, Panagiotopoulos S, Tipping P. Super High Flux Hemofiltration: A new technique for cytokine removal. Intensive Care Med 2002; 28: 651-655
   16. De Vriese AS, Francis AC, Philippe JJ, et al. (1999) Cytokine removal during continuous hemofiltration in septic patients. J Am Soc Nephrol 10:846-853
   17. Kellum JA, Johnson JP, Kramer D, Pavelsky P, Brady JJ, Pinsly MR. Diffusive vs convective therapy: effects on mediators of inflammation in patient with severe systemic inflammatory response syndrome. Crit Care Med 1998; 26(12): 1995-2000.
   18. Opal SM. Hemofiltration-absorption systems for the treatment of experimental sepsis: is it possible to remove the "evil humors" responsible for septic shock? Crit Care Med 2000; 28(5): 1681-1682.
   19. Bellomo R, Baldwin I, Ronco C. High-volume hemofiltration. Current Opinion in Critical Care 2000; 6: 442-445
   20. Cole L, Bellomo R, Journois D, Davenport P, Baldwin I, Tipping P. High volume hemofiltration in human septic shock. Intensive Care Med 2001; 27: 978-986
   21. The ACCP/SCCM Consensus conference committee: Bone RC, Balk RA, Cerra FB, Dellinger RP,Fein AM, Knaus WA, Schein RMH, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Chest 1992; 101:1644-55.
   22. Bach LA, Sharpe K, Sample size for clinical and biological research. Aust NZ J Med 1989; 19: 64-67
   23. Ronco, C; Brendolan, A; Lonnemann, G; Bellomo, R; Piccinni, P; Digito, A; Dan, M; Irone, M; LaGreca, G; Inguaggiato, P; Maggiore, U; DeNitti, C Wratten, M; Ricci, Z &Tetta,c. (2002) Apiolt study of coupled filtration with adsorption in septic shock. Critical Care Medicine, June 2002 Vol 30 No 6 p.p. 1250-1256

ELIGIBILITY:
Inclusion Criteria:

* All patients who fulfil the consensus criteria for sepsis (21) and recently proposed criteria for severe ARF (1) are eligible for the study.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients who are pregnant or breastfeeding
* Patients with a known allergy to polyamide
* Patients expected to die within 24 hours
* Patients in whom there are limitations on the intensity of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2006-06; Study Completion 2006-11

PRIMARY OUTCOMES:
The primary outcome measure for this study is the relative change in plasma IL-6 levels.

SECONDARY OUTCOMES:
The secondary outcome is the clearance and the absolute change in the levels of IL-6 and other cytokines.
The other secondary outcome is the change in noradrenaline dose required to maintain baseline mean blood pressure (typically 70 mmHg)
change in the levels of other cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, MD, FRACP, Principal Investigator — Austin Health
Locations (1):
- Austin Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Haase M, Bellomo R, Baldwin I, Haase-Fielitz A, Fealy N, Davenport P, Morgera S, Goehl H, Storr M, Boyce N, Neumayer HH. Hemodialysis membrane with a high-molecular-weight cutoff and cytokine levels in sepsis complicated by acute renal failure: a phase 1 randomized trial. Am J Kidney Dis. 2007 Aug;50(2):296-304. doi: 10.1053/j.ajkd.2007.05.003. PMID 17660031
- [Derived] Haase M, Bellomo R, Baldwin I, Haase-Fielitz A, Fealy N, Morgera S, Goehl H, Storr M, Boyce N, Neumayer HH. Beta2-microglobulin removal and plasma albumin levels with high cut-off hemodialysis. Int J Artif Organs. 2007 May;30(5):385-92. doi: 10.1177/039139880703000505. PMID 17551901